CLINICAL TRIAL: NCT01434134
Title: Prevention of Cardiac Dysfunction During Adjuvant Breast Cancer Therapy: A Randomized, Placebo-controlled, 2x2 Factorial, Double Blind Trial of Candesartan and Metoprolol
Brief Title: Prevention of Cardiac Dysfunction During Adjuvant Breast Cancer Therapy
Acronym: PRADA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other); Norwegian Cancer Society (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Torbjorn Omland, Professor of Medicine, University Hospital, Akershus
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2709001/90005
Record Dates: First submitted 2011-09-05; First posted 2011-09-14 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer; Heart Failure
Keywords: Anthracyclines; Trastuzumab
MeSH Terms: conditions — Breast Neoplasms; Heart Failure | interventions — Metoprolol; candesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Metoprolol (Experimental): Tablet, target dose 100 mg once daily
  Interventions: Drug: Metoprolol
- Placebo for Metoprolol (Placebo Comparator): Tablet, target dose 100 mg once daily
  Interventions: Drug: Placebo
- Candesartan (Experimental): Tablet, target dose 32 mg once daily
  Interventions: Drug: Candesartan
- Placebo for Candesartan (Placebo Comparator): Tablet, target dose 32 mg once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoprolol — Tablet, target dose 100 mg once daily
  Arms: Metoprolol
Drug: Placebo — Tablet, target dose 100 mg once daily
  Arms: Placebo for Metoprolol
Drug: Candesartan — Tablet, target dose 32 mg once daily
  Arms: Candesartan
Drug: Placebo — Tablet, 32 mg once daily
  Arms: Placebo for Candesartan

SUMMARY:
Women treated for breast cancer are at increased risk for cardiovascular disease, including heart failure. In this study, by using magnetic resonance imaging (MRI), the investigators want to assess if heart failure medications such as beta blockers and angiotensin receptor blockers can prevent cardiac dysfunction during early breast cancer therapy.

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignancies in women. Recent progress in the detection and treatment of breast cancer has resulted in survival gains, but a consequence of therapeutic advances is an increasing number of long-term survivors who may be at risk for development of cardiovascular disease. Several studies suggest that women treated for breast cancer may be at increased risk for cardiovascular disease, the probable causes being multi-factorial. Importantly, therapies for breast cancer, including radiotherapy, anti-HER-2 regimens and certain chemotherapeutic regimens, may increase the risk of subsequent cardiovascular disease, including atherosclerotic disease, left ventricular dysfunction, and heart failure.

In the current study we propose to undertake a randomized, placebo-controlled, 2x2 factorial, double-blind trial to assess whether left ventricular dysfunction and/or injury is preventable, completely or partly, by the concomitant administration of the angiotensin receptor blocker (ARB), candesartan, and the beta blocker, metoprolol, during postoperative chemotherapy and radiotherapy.

The proposed study addresses an important clinical problem in a large patient group. Thus, the possibility of preventing cardiovascular side effects of contemporary therapy for breast cancer is important both clinically and scientifically.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-70 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Serum creatinine < 140 μmol/L or estimated creatinine clearance > 60 ml/min (using the modification of diet and renal disease (MDRD) formula)
* Systolic blood pressure >= 110 mgHg and < 170 mmHg
* LVEF >= 50%

Exclusion Criteria:

* Hypotension, defined as systolic blood pressure < 110 mmHg
* Bradycardia, defined as heart rate < 50 b.p.m.
* Prior anthracycline chemotherapy regimen
* Prior malignancy requiring chemotherapy or radiotherapy
* Symptomatic heart failure
* Systolic dysfunction (LVEF < 50%)
* Clinically significant coronary artery disease, valvular heart disease, significant arrhythmias, or conduction delays.
* Uncontrolled arterial hypertension defined as systolic blood pressure > 170 mm Hg
* Treatment with ACEI, ARB or beta-blocker within the last 4 weeks prior to study start
* Intolerance to ACEI, ARB or beta-blocker
* Uncontrolled concomitant serious illness
* Pregnancy or breastfeeding
* Active abuse of drugs or alcohol
* Suspected poor compliance
* Inability to tolerate the MRI scanning protocol

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction, as assessed by cardiac MRI | Baseline and end of study (up to 72 weeks)

SECONDARY OUTCOMES:
Change in contrast enhancement by MRI | Baseline and approximately 4 weeks
Change in left 2D global strain, as assessed by echocardiography | Baseline and end of study (up to 72 weeks)
Incidence of clinical of heart failure or objective left ventricular dysfunction | Up to 72 weeks
  Left ventricular dysfunction defined as ejection fraction < 55% by cardiac MRI
Change in biochemical markers of cardiac injury, i.e. hs-cTnT | Baseline and end of study (up to 72 weeks)
Change in left ventricular diastolic function, as assessed by echocardiography | Baseline and end of study (up to 72 weeks)
  Diastolic function assessed by e/e'
Change in biochemical markers of cardiac function, i.e. NT-proBNP | Baseline and end of study (up to 72 weeks)
Change in contrast enhancement, as assessed by cardiac MRI | Baseline and end of study (up to 72 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Stein Vaaler, Study Director — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

REFERENCES:
- [Derived] Mecinaj A, Gulati G, Ree AH, Gravdehaug B, Rosjo H, Steine K, Wisloff T, Geisler J, Omland T, Heck SL. Impact of the ESC Cardio-Oncology Guidelines Biomarker Criteria on Incidence of Cancer Therapy-Related Cardiac Dysfunction. JACC CardioOncol. 2024 Jan 16;6(1):83-95. doi: 10.1016/j.jaccao.2023.10.008. eCollection 2024 Feb. PMID 38510299
- [Derived] Heck SL, Mecinaj A, Ree AH, Hoffmann P, Schulz-Menger J, Fagerland MW, Gravdehaug B, Rosjo H, Steine K, Geisler J, Gulati G, Omland T. Prevention of Cardiac Dysfunction During Adjuvant Breast Cancer Therapy (PRADA): Extended Follow-Up of a 2x2 Factorial, Randomized, Placebo-Controlled, Double-Blind Clinical Trial of Candesartan and Metoprolol. Circulation. 2021 Jun 22;143(25):2431-2440. doi: 10.1161/CIRCULATIONAHA.121.054698. Epub 2021 May 16. PMID 33993702
- [Derived] Gulati G, Heck SL, Rosjo H, Ree AH, Hoffmann P, Hagve TA, Norseth J, Gravdehaug B, Steine K, Geisler J, Omland T. Neurohormonal Blockade and Circulating Cardiovascular Biomarkers During Anthracycline Therapy in Breast Cancer Patients: Results From the PRADA (Prevention of Cardiac Dysfunction During Adjuvant Breast Cancer Therapy) Study. J Am Heart Assoc. 2017 Nov 8;6(11):e006513. doi: 10.1161/JAHA.117.006513. PMID 29118031
- [Derived] Heck SL, Gulati G, Ree AH, Schulz-Menger J, Gravdehaug B, Rosjo H, Steine K, Bratland A, Hoffmann P, Geisler J, Omland T. Rationale and design of the prevention of cardiac dysfunction during an Adjuvant Breast Cancer Therapy (PRADA) Trial. Cardiology. 2012;123(4):240-7. doi: 10.1159/000343622. Epub 2012 Nov 30. PMID 23207160